CLINICAL TRIAL: NCT06389435
Title: ROCKETS: RObotic-assisted Versus Conventional Knee Endoprosthetic Techniques in a Randomized, Multicenter, Preference-tolerant Study
Brief Title: RObotic-assisted Versus Conventional Knee Endoprosthetic Techniques
Acronym: ROCKETS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other); Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Olof Skoldenberg, Professor, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024DS; Knee (Other: Danderyds sjukhus)
Record Dates: First submitted 2024-04-04; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Knee Arthroplasty, Total; Robotic-assisted; Osteoarthritis of the Knee
Keywords: Knee arthroplasty; Robotic assisted; Osteoartritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RTKR (Experimental): Robotic assisted total knee replacement (RTKR)
  Interventions: Procedure: Patients will be randomized to undergo TKR or RTKR
- TKR (Active Comparator): Standard total knee replacement (TKR)
  Interventions: Procedure: Patients will be randomized to undergo TKR or RTKR

INTERVENTIONS:
Procedure: Patients will be randomized to undergo TKR or RTKR — Total knee replacement (control group)

SUMMARY:
Rationale for conducting the study:

The study aims to systematically evaluate the clinical and economic impacts of Robotic-Assisted Total Knee Replacement (RTKR) compared to conventional Total Knee Replacement (TKR). It focuses on the potential benefits of RTKR, including improved precision in surgery, potentially leading to better patient outcomes and reduced healthcare costs. Our primary endpoint is the Forgotten Joint Score (FJS), aimed at measuring patients awareness of their knee joint in everyday life, indicating the success of the knee replacement surgery in restoring natural joint function. Secondary endpoints include patient-reported outcome measures (PROMs), patient activity levels, the accuracy of implant positioning on x-ray, and the incidence of adverse events.

Study design:

Multicentre,, preference-tolerant, randomized, controlled, superiority trial with two treatment arms that compares the outcomes of RTKR with traditional TKR techniques.

Study population:

Adult patients aged 18 years and older who are eligible for TKR as per local guidelines and who have given informed consent to participate in the study.

Number of patients:

400

Inclusion criteria:

Patients must be adults aged 18 years and older, eligible for TKR according to local guidelines, and willing to participate in the study.

Exclusion criteria:

Patients with extreme malalignment requiring special implants or techniques, patients unfit for surgery due to medical reasons, and those deemed unsuitable to participate in the study for other reasons.

Primary outcome variables:

The Forgotten Joint Score (FJS) at 2 years after surgery

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older.
* Eligible for TKR according to local guidelines and routines.
* Willingness to participate in the study.

Exclusion Criteria:

* Patients with extreme malalignment necessitating special implants or techniques.
* Patients unfit for surgery due to other medical reasons.
* Patients who, for other reason such as alcohol or substance abuse, is deemed unsuitable to participate in the study.
* Patients who, for other reasons can't fulfill the required patient recorded outcome measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The Forgotten Joint Score (FJS) | 24 months post surgery
  The primary outcome measurement will be the Forgotten Joint Score (FJS), measured at 24 months post-surgery. The FJS evaluates the patient's ability to 'forget' the artificial joint in their daily life. This scale ranges from 0 to 100, where 0 represents the maximum joint awareness and 100 represents complete joint unawareness, indicating that the patient does not perceive the joint during daily activities. Higher scores indicate a better outcome, reflecting the success of the knee replacement surgery in restoring natural joint function such that the joint feels like a natural part of the body.

SECONDARY OUTCOMES:
KOOS | preop, 6 weeks, 12 and 24 months post surgery
  The secondary outcome measure will include the Knee Injury and Osteoarthritis Outcome Score (KOOS). The KOOS is designed to assess patients' opinions about their knee and associated problems. The score comprises five separately scored subscales: Pain, Other Symptoms, Function in Daily Living (ADL), Function in Sport and Recreation (Sport/Rec), and Knee-Related Quality of Life (QOL). Each subscale is scored from 0 to 100, where 0 represents extreme knee problems and 100 represents no knee problems. Higher scores indicate a better outcome, reflecting fewer symptoms and higher levels of knee function in daily and recreational activities.
ADLS knee instability | 6 weeks, 12 and 24 months post-operation.
  The self reported Activities of Daily Living Scale of the Knee Outcome Survey (ADLS) where participants will rate, over the previous 1-2 days, the degree to which slipping/partial giving way (item 1) and buckling/full giving way (item 2) of each knee affected daily activity graded from 0 (no) to 6 (severe impact on daily living)
The Forgotten Joint Score (FJS) | 6 weeks and 12 months post surgery
  A secondary outcome measurement will be the Forgotten Joint Score (FJS), measured preoperatively, and at 6 weeks and 12 months post-surgery. The FJS evaluates the patient's ability to 'forget' the artificial joint in their daily life. This scale ranges from 0 to 100, where 0 represents the maximum joint awareness and 100 represents complete joint unawareness, indicating that the patient does not perceive the joint during daily activities. Higher scores indicate a better outcome, reflecting the success of the knee replacement surgery in restoring natural joint function such that the joint feels like a natural part of the body.
EQ-5D | 6 weeks, 12 and 24 months post surgery
  A secondary outcome measure will be the European Quality of Life-5 Dimensions (EQ-5D). The EQ-5D is a standardized instrument used to measure health-related quality of life that can be utilized in a wide range of health conditions and treatments. This tool includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels: no problems, some problems, and extreme problems. The EQ-5D index is calculated by applying a formula that attaches values to each of the levels in each dimension. This index can range from -0.594 to 1.0, where 1.0 indicates the best health state, 0 represents death, and negative values represent health states perceived as worse than death.
Knee alignment | 6 weeks post surgery
  Knee alignment measured with long standing x-ray
Adverse events | up to 24 months post surgery
  Adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Danderyds Sjukhus, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No